CLINICAL TRIAL: NCT00569036
Title: A Phase I Multiple Ascending Dose Study of BMS-754807 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Multiple Dose Study In Cancer Patients: Safety and Tolerability of BMS-754807 in Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA191-002
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Neoplasms; Solid Tumors; Metastases
Keywords: Advanced or Metastatic Solid Tumors or Neoplasms
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — BMS 754807

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-754807 (Experimental): Single arm, multiple-ascending dose escalation study
  Interventions: Drug: BMS-754807

INTERVENTIONS:
Drug: BMS-754807 — Tablets, Oral, Dose Cohorts: 4mg, 10mg, 20mg, 30mg, 50mg, 70mg, 100mg, 130mg, 160mg, 200mg, Once Daily, Until disease progression, unacceptable toxicity or at the subject's request
  Other Names: IGF-IR

SUMMARY:
This is a Phase 1 dose escalation study to determine the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary anti-tumor activity of BMS-754807 in patients with advanced or metastatic solid tumors. In addition, the study is expected to identify the recommended dose or dose range of BMS-754807 for Phase 2 studies

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced or metastatic solid tumors for whom the standard of care is ineffective or inappropriate
* ECOG performance status 0-1
* at least 4 weeks between surgery or last dose prior anti-cancer therapy

Exclusion Criteria:

* symptomatic brain metastases
* any disorder or dysregulation of glucose homeostasis {e.g. diabetes)
* uncontrolled or significant cardiovascular disease
* inadequate bone marrow, liver or kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety - Toxicities will be evaluated according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 3 | Continuous assessment throughout the duration of the trial

SECONDARY OUTCOMES:
Pharmacokinetics | assessed during the first 4 weeks of the study
Pharmacodynamics | assessed during the first 4 weeks of the study
Metabolic measures | assessed during the first 4 weeks of the study
ECG | assessed during the first 4 weeks of the study
Efficacy Measures | assessed every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- Australia (5):
  - Local Institution, East Melbourne, Victoria
  - Local Institution, Footscray, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Parkville, Victoria
  - Local Institution, Nedlands, Western Australia

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx